CLINICAL TRIAL: NCT01157052
Title: Oxaliplatin Pharmacokinetics With and Without Ca2+/MG2+ Infusion in Colorectal Cancer Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25408
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Neoplasms, Colorectal; Colorectal Cancer; Colorectal Carcinoma
Keywords: magnesium; calcium; adverse effects; kinetics, drug
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Calcium; Magnesium; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ca2+/Mg2+ pre & post cycle 1 (Active Comparator): Arm A:Ca2+/Mg2+: Ca++gluconate 1gr & Mg++sulfate 1g given IV pre & post cycle 1
  Interventions: Other: (supplement) Calcium and Magnesium
- Ca2+/Mg2+pre & post cycle 2 (Active Comparator): Arm B:Ca2+/Mg2+: Ca++gluconate 1gr & Mg++sulfate 1g given IV pre & post cycle 2
  Interventions: Other: (supplement) Calcium and Magnesium

INTERVENTIONS:
Other: (supplement) Calcium and Magnesium — FOLFOX 6: Oxaliplatin (Eloxatin®): 100mg/m2 x 2hrs IV with 250ml of dextrose 5%; leucovorin 200mg/m2 with oxaliplatin; then IV bolus of 5FU 400mg/m2 and 5FU 2400mg/m2 in a 46 hr continuous IV. Each cycle is 14 days, approximately 8-12 cycles planned.
  XELOX: Oxaliplatin 130mg/m2 x 2hrs IV in 250ml of dextrose 5% on day 1; plus oral capecitabine 1000mg/m2 bid on days 1-15 3 wk cycles.
  Ca2+/Mg2: Ca++gluconate 1gr & Mg++sulfate 1g given IV pre & post cycle 1 (Arm A) or cycle 2 (Arm B)
  Other Names: oxaliplatin= eloxatin, Capecitabine=Xeloda

SUMMARY:
The investigators hypothesize that Ca2+/MG2+ infusions will not have a significant effect on oxaliplatin pharmacokinetics.

DETAILED DESCRIPTION:
This is a clinical pharmacology prospective non-randomized trial to determine oxaliplatin pharmacokinetics in the presence and absence of calcium and magnesium supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have Metastatic Colorectal Cancer (stage IV)
* Patients who were treated with 5FU and leucovorin in the adjuvant setting or with 5FU and leucovorin (LV)or/and FOLFIRI regimen for metastatic setting may be eligible for this trial.
* Patients must be ≥ 18 years
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Patients must have adequate renal function of creatinine < 1.5mg/dl and a creatinine clearance > 45ml/min. Patients must have adequate hepatic function with a bilirubin > 1.5 mg/dl and AST (normal range 0-14/L) and ALT (normal range 0-49 U/L) in the absence of liver metastasis or </= 5X the upper limit of normal of AST and ALT in the presence of liver metastasis.
* Patients must have adequate bone marrow function with absolute neutrophil count(ANC)≥ 1,500/цl and platelets ≥ 100,000/цl and a hemoglobin ≥ 10g/d.
* Patients must be willing and able to comply with the study protocol for the study duration and patients must give written informed consent prior to any study-specific screening procedures with the understanding that the patient may withdraw consent at any time without prejudice.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment. Also,women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation. The investigator is requested to advise the patient how to achieve an adequate contraception.
* Life expectancy longer that 6 months

Exclusion Criteria:

* Patients who have received oxaliplatin previously
* Patients with known peripheral neuropathy ≥ grade 2 according to the WHO scale
* Patients who have tested positive for HIV
* Patients with other significant medical, psychiatric disorders tha, in the opinion of the investigator, will exclude the patient from the study for compliance of safety reasons.
* Patients who cannot swallow
* History of known allergy to oxaliplatin or other platinum compounds,to 5-FU, to LV, or to any ingredients in the formulations or the containers
* Participation in another clinical trial with any investigational drug within 30 days prior to study screening
* Pernicious anemia or other megaloblastic anemia with vitamin B12 deficiency
* Patient with concomitant treatment with drugs/ingredients reported to have a potential activity to prevent peripheral sensory neuropathy (PSN)
* Patients who haven't successfully completed local therapy for previously treated CNS metastases & who haven't been discontinued with corticosteroid for >4kws before starting chemotherapy. Patients with asymptomatic brain mets who have no evidence of midline shift on CT/MRI may be enrolled without initiation of local therapy for the CNS mets. Repeat scan must be performed < 4wks to ensure no progression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to determine potential pharmacokinetic interactions between oxaliplatin and calcium and magnesium. | Post cycle 2 and 3

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sawyer, MD, Study Chair — Alberta Health services
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada